CLINICAL TRIAL: NCT02840825
Title: Biochip for HCMV Detection in Breast Milk From Lactating Women of Preterm Infants Less Than 33 Weeks
Brief Title: Biochip for HCMV Detection in Breast Milk
Acronym: VIRUMILK
Status: Terminated | Type: Observational
Why Stopped: Technical issues with microchip
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: API/2015/63
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Cytomegalovirus Infections; Breast Feeding; Premature Birth of Newborn
MeSH Terms: conditions — Cytomegalovirus Infections; Breast Feeding; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — breastmilk
Oversight: Data Monitoring Committee: No

SUMMARY:
Human cytomegalovirus (HCMV) is the leading cause of neonatal viral infection and can have a significant impact on the neurosensory development of newborns and especially preterm infants. HCMV infection may result from maternal-fetal transmission during pregnancy or postnatal transmission. While congenital HCMV infection affects about 2-5% of very preterm infants, the risk of postnatal infection, particularly through breast milk, is much higher in this population (prevalence of about 20%). Many learned societies wonder about the interest to inactivate HCMV (by freezing or pasteurization) in breast milk in order to reduce or eliminate contamination of these children. However, freezing is relatively inefficient to reduce contamination and pasteurization drastically alters the nutritional quality of the milk. Therefore, a systematic preventive treatment of breast milk for very preterm infants is not currently recommended. An alternative approach could consist in detecting HCMV in breast milk to target at-risk situations. This detection can be performed by PCR but its cost and the time required to obtain the result prohibits its use for a mass detection. Currently, viral status of breast milk is not explored in practice and, depending on the health centers, breastfeeding is continued as such or milk is systematically inactivated.The main objective of VIRUMILK is to study the feasibility of the CMV detection in breast milk from lactating mothers with a biochip.The ultimate goal is to prevent postnatal HCMV infection of preterm newborns less than 33 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Lactating women (> 18 years)
* Mothers with infants less than 33 weeks hospitalized in intensive care infant / neonatal the University Hospital of Besancon.
* No opposition mothers.
* Join a French social security or receiving such a scheme.
* Subjects who received medical care during pregnancy.

Exclusion Criteria:

* Legal incapacity or limited legal capacity.
* Topics without health insurance.
* Topics being in the disqualification of another study or under the "national register of volunteers."

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be proposed to mothers meeting the criteria described in part "Eligibility criteria" during an investigators' visit of the newborn infant in the Department of Neonatal Medicine of the Besancon University Hospital. They will then receive information on the study. The practitioner responsible for the study will also collect non-opposition of mothers.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
optical detection of HCMV specifically captured on the biochip with respect to the reference (PCR) technique. | Within 4 days after receiving the breast milk sample

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Thiriez, MD, PhD, Principal Investigator — Centre hospitalier régional universitaire de Besançon
Locations (1):
- CHRU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided